CLINICAL TRIAL: NCT04124939
Title: A Randomized Clinical Trial of 100 Units of Intradetrusor Onabotulinum Toxin A for Refractory Overactive Bladder - Is 10 Injections Less Painful Than 20 Injections?
Brief Title: Is 10 Injections of Bladder Botox Less Painful Than 20 Injections?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00059454
Record Dates: First submitted 2019-10-10; First posted 2019-10-14 (Actual); Results first posted 2023-10-13 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2022-08

CONDITIONS: Overactive Bladder
Keywords: Overactive Bladder; Botox/OnabotulinumtoxinA; Pain; OAB; Non-neurogenic Overactive bladder
MeSH Terms: conditions — Urinary Bladder, Overactive; Pain | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 10 Botox Injections (Active Comparator): 100 units of Botox® (onabotulinumtoxinA) will be combined with 10 cc of sterile saline for the purpose of 10 injections. The bladder will be instilled with 2% lidocaine solution through a catheter for at least 5 minutes prior to the procedure. Cystoscopy with either a rigid or flexible cystoscope (per surgeon preference) will be performed using sterile technique. The Botox® will be injected in a grid like pattern avoiding the trigone.
  Interventions: Drug: OnabotulinumtoxinA 100 Units
- 20 Botox Injections (Active Comparator): 100 units of Botox® (onabotulinumtoxinA) will be combined with 20 cc of sterile saline for the purpose of 20 injections. The bladder will be instilled with 2% lidocaine solution through a catheter for at least 5 minutes prior to the procedure. Cystoscopy with either a rigid or flexible cystoscope (per surgeon preference) will be performed using sterile technique. The Botox® will be injected in a grid like pattern avoiding the trigone.
  Interventions: Drug: OnabotulinumtoxinA 100 Units

INTERVENTIONS:
Drug: OnabotulinumtoxinA 100 Units — BOTOX for injection is an acetylcholine release inhibitor and a neuromuscular blocking agent indicated for:
  • Treatment of overactive bladder (OAB) with symptoms of urge urinary incontinence, urgency, and frequency, in adults who have an inadequate response to or are intolerant of an anticholinergic medication.
  Other Names: BOTOX

SUMMARY:
The purpose of this research study is to help determine if 10 injections of Botox ® 100 units is less painful than 20 injections of Botox ® 100 units based on effectiveness in reducing urge incontinence episodes. Study will also be assessed for the pain of procedure and adverse outcomes of 20 injections versus 10 injections.

DETAILED DESCRIPTION:
This study is a randomized clinical trial to assess whether or not 10 injections of 100 units of intradetrusor Botox® toxin is perceived as less painful compared to 20 injections of 100 units of intradetrusor Botox® toxin for the treatment of refractory overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* At least 18 years of age
* Have already decided to undergo intradetrusor Botox® injections for treatment of refractory overactive bladder.
* Able and willing to learn clean intermittent catheterization (or care provider is willing and able to perform intermittent catheterization).
* Understands and is willing to undergo follow up and complete questionnaires as described in this protocol
* Able to give informed consent

Exclusion Criteria:

* Male gender
* Neurological conditions (Examples: Cerebral vascular accident within 6 months prior to treatment, Parkinson's disease, Multiple Sclerosis, and Spina Bifida).
* Acute urinary tract infection
* Treatment with Botox® toxin for other conditions
* Allergy to Botox® toxin
* Hematuria that has not been worked up
* Known bladder malignancy
* Previous history of bladder augmentation
* Currently pregnant (with no plans to become pregnant within 6 months of enrollment) or breastfeeding
* Currently taking aminoglycoside antibiotics
* Post-void residual (PVR) >150 cc (measured by bladder scan or by catheterization) prior to enrollment
* History of chronic pain or pain syndromes

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 41 (Actual)
Dates: Start 2019-11-10 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2023-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Matthews, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Urology clinic locations at Wake Forest Baptist Medical Center, Greensboro, North Carolina
  - Urology clinic locations at Wake Forest Baptist Medical Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 154 patients found eligible for study trial participation. 89 of 154 did not meet the inclusion criteria, 14 declined participation, and 10 patients with other reasons did not participate. Total 41 patients participated with 21 in 10 injections arm and 20 in 20 injections arm.21 patients of 10 injections arm and 19 of 20 injection arm were accounted in study analysis.
Groups:
- 10 Botox Injections: 100 units of Botox® (onabotulinumtoxinA) will be combined with 10 cc of sterile saline for the purpose of 10 injections. The bladder will be instilled with 2% lidocaine solution through a catheter for at least 5 minutes prior to the procedure. Cystoscopy with either a rigid or flexible cystoscope (per surgeon preference) will be performed using sterile technique. The Botox® will be injected in a grid like pattern avoiding the trigone.
  OnabotulinumtoxinA 100 UNT: BOTOX for injection is an acetylcholine release inhibitor and a neuromuscular blocking agent indicated for:
  • Treatment of overactive bladder (OAB) with symptoms of urge urinary incontinence, urgency, and frequency, in adults who have an inadequate response to or are intolerant of an anticholinergic medication.
- 20 Botox Injections: 100 units of Botox® (onabotulinumtoxinA) will be combined with 20 cc of sterile saline for the purpose of 20 injections. The bladder will be instilled with 2% lidocaine solution through a catheter for at least 5 minutes prior to the procedure. Cystoscopy with either a rigid or flexible cystoscope (per surgeon preference) will be performed using sterile technique. The Botox® will be injected in a grid like pattern avoiding the trigone.
  OnabotulinumtoxinA 100 UNT: BOTOX for injection is an acetylcholine release inhibitor and a neuromuscular blocking agent indicated for:
  • Treatment of overactive bladder (OAB) with symptoms of urge urinary incontinence, urgency, and frequency, in adults who have an inadequate response to or are intolerant of an anticholinergic medication.
Period: Overall Study
Arm/Group | 10 Botox Injections | 20 Botox Injections
Started | 21 | 20
Completed | 20 | 17
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 Botox Injections | 20 Botox Injections | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.28 (8.97) | 67.67 (9.10) | 69.67 (9.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: Numeric Pain Rating Scale (NPRS)
Description: The patients will rate their level of pain from 0 as no pain to 10 as a severe pain immediately following the completion of bladder injections by selecting a whole number from 0 to 10 that represents their level of pain during the procedure.
Time Frame: Post Procedure Day 1
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | 10 Botox Injections | 20 Botox Injections
Number analyzed (Participants) | 21 | 19
score on a scale | 4 [1.5 to 5] | 3 [1 to 4]

2. Secondary Outcome: Difference in Mean Urge Incontinence Episodes
Description: The mean urge incontinence episodes which will be calculated by averaging the amount of urge urinary incontinence episodes over 3 days as recorded in a bladder diary at week 12 after the procedure
Time Frame: Week 12 after procedure
Measure: Mean (Inter-Quartile Range); unit: Number of Urinary Leaks in 24 HRS
Arm/Group | 10 Botox Injections | 20 Botox Injections
Number analyzed (Participants) | 20 | 17
Number of Urinary Leaks in 24 HRS | 1.64 [1 to 1.82] | 1.35 [0 to 2]

3. Secondary Outcome: Over Active Bladder (OAB) Questionnaire Short Form Scores - Symptoms
Description: Secondary endpoints to be assessed as OAB symptoms using Overactive Bladder Questionnaire Short Form (OABq-SF) at baseline, 2 weeks and 12 week post-procedure. 0 - to 100-point scale, with lower scores indicating greater effect, i.e., worse Quality of Life
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 10 Botox Injections | 20 Botox Injections
Number analyzed (Participants) | 21 | 19
score on a scale | 29.67 (5.43) | 25.89 (7.45)

4. Secondary Outcome: Over Active Bladder (OAB) Questionnaire Short Form Scores - Symptoms
Description: as for outcome 3
Time Frame: 2 weeks post procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 10 Botox Injections | 20 Botox Injections
Number analyzed (Participants) | 21 | 17
score on a scale | 17.1 (7.21) | 17.0 (17.83)

5. Secondary Outcome: Over Active Bladder (OAB) Questionnaire Short Form Scores - Symptoms
Description: as for outcome 3
Time Frame: 12 weeks post procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 10 Botox Injections | 20 Botox Injections
Number analyzed (Participants) | 20 | 17
score on a scale | 15.53 (6.18) | 16.41 (6.48)

6. Secondary Outcome: Over Active Bladder (OAB) Questionnaire Short Form Scores - Health Related Quality of Life
Description: Secondary endpoints to be assessed as OAB symptoms using Overactive Bladder Questionnaire Short Form (OABq-SF) at baseline, 2 weeks and 12 week post-procedure. 13 items to assess health Related Quality of Life (HRQOL). Total range 0 to 100. A higher score on the HRQOL scale indicates a better HRQO.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 10 Botox Injections | 20 Botox Injections
Number analyzed (Participants) | 21 | 19
score on a scale | 56.04 (13.46) | 47.94 (20.36)

7. Secondary Outcome: Over Active Bladder (OAB) Questionnaire Short Form - Health Related Quality of Life
Description: as for outcome 6
Time Frame: 2 weeks post procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 10 Botox Injections | 20 Botox Injections
Number analyzed (Participants) | 21 | 17
score on a scale | 28.71 (14.26) | 23.63 (14.04)

8. Secondary Outcome: Over Active Bladder (OAB) Questionnaire Short Form - Health Related Quality of Life
Description: as for outcome 6
Time Frame: 12 weeks post procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 10 Botox Injections | 20 Botox Injections
Number analyzed (Participants) | 20 | 17
score on a scale | 27.74 (12.92) | 27.00 (11.20)

9. Secondary Outcome: Post-Void Residual (PVR)
Description: PVR using bladder scanner evaluates the post void residual in the bladder.
Time Frame: 2 weeks post procedure
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | 10 Botox Injections | 20 Botox Injections
Number analyzed (Participants) | 21 | 17
ml | 93.87 (79.37) | 71.93 (89.62)

10. Secondary Outcome: Post-Void Residual (PVR)
Description: PVR using bladder scanner evaluates the post void residual in the bladder.
Time Frame: 12 weeks post procedure
Measure: Mean (Inter-Quartile Range); unit: ml
Arm/Group | 10 Botox Injections | 20 Botox Injections
Number analyzed (Participants) | 20 | 17
ml | 17.5 [0 to 91] | 61 [0 to 125]

ADVERSE EVENTS:
Time Frame: 12 Weeks
Arm/Group | 10 Botox Injections | 20 Botox Injections
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 4/21 | 5/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 Botox Injections (N=21) | 20 Botox Injections (N=20)
Urinary Tract Infection (Renal and urinary disorders) | 4 (4) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/39/NCT04124939/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-31): https://cdn.clinicaltrials.gov/large-docs/39/NCT04124939/SAP_001.pdf
  • Informed Consent Form (2022-07-12): https://cdn.clinicaltrials.gov/large-docs/39/NCT04124939/ICF_002.pdf